CLINICAL TRIAL: NCT04752618
Title: Treating Maternal PTSD to Enhance and Reduce Maltreatment Recidivism: Safe Mothers, Safe Children
Brief Title: Safe Mothers, Safe Children Initiative
Acronym: SMSC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-FY2021-5220
Record Dates: First submitted 2021-01-29; First posted 2021-02-12 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-11

CONDITIONS: PTSD; Depression; Child Maltreatment
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression

STUDY DESIGN:
Intervention Model Description: P-STAIR vs Supportive Counseling
Who Masked: Outcomes Assessor
Masking Description: Assessors and preventive case planners are blind to treatment arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- P-STAIR (Experimental): Participants will receive 23 weekly individual treatment sessions. Each session will last one hour. P-STAIR is a combination of STAIR and PCIT. STAIR focuses on reduction of PTSD symptoms through enhancement of emotion regulation skills. PCIT focuses on the reduction of negative parenting skills and the increase of positive parenting skills.
  Interventions: Behavioral: P-STAIR
- Supportive Counseling (Active Comparator): Participants will receive 23 weekly individual treatment sessions. Each session will last one hour. Supportive counseling has been modified to permit non-trauma discussion of parenting problems. Each session is client-directed and clinicians take an unconditionally supportive role.
  Interventions: Behavioral: Supportive Counseling

INTERVENTIONS:
Behavioral: P-STAIR — PCIT+ STAIR
  Arms: P-STAIR
Behavioral: Supportive Counseling — Non-trauma focused psychotherapy
  Arms: Supportive Counseling

SUMMARY:
The purpose of this study is to assess the efficacy of the combined interventions, Skills Training in Affective and Interpersonal Regulation (STAIR) and Parent-Child Interaction Therapy (PCIT) or P-STAIR, for treating maternal PTSD and reducing maltreatment recidivism.

DETAILED DESCRIPTION:
This study is a two-arm randomized controlled trial (RCT): P-STAIR (23 sessions) vs. supportive counseling (SC) (23 sessions). Eligible cases are randomized to P-STAIR and SC in a 1:1 ratio. Participants will be mothers receiving family preservation services (FPS), with a child in the age range of 1-10 years old, and PTSD (with/without depression). Symptom progress will be measured at pre-treatment, two in-treatment assessments (9 weeks and 16 weeks), post-treatment, and at a 6-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Receiving preventive services at the time of the consent session to participate in the study
* Meeting a severity score of 28 or higher OR probable DSM-5 diagnostic criteria for PTSD (PDS-5)
* Having 1-10-year-old child
* Being the legal guardian for the child with physical and legal custody
* Being able to read, write, and speak English or Spanish

Exclusion Criteria:

* Having suicidal ideation present in the past month prior to pre-assessment or reports of a suicide attempt in the past year (SCID-5)
* Meeting a diagnosis of severe substance or alcohol use disorder (≥ 6 symptoms on SCID) AND not in early remission (≥3 months without meeting any substance or alcohol use disorder criteria (except craving)
* Having current or active symptoms of psychosis in the past month
* Having a disability affecting communication, such as deafness
* Having an index child with a developmental condition that impedes cognitive and/or physical functioning, e.g. autism
* Having an index child with current symptoms or diagnosis of psychosis as defined by the DSM-5 in the past 3 months
* Experiencing current or history of intimate partner violence (IPV) or family violence:

If there is a history of IPV/family violence and the relationship is no longer active, the relationship must have ended for at least ninety days with no intention of restarting; If there is a history of IPV/family violence, but the relationship is ongoing, there must not have been an IPV/family violence event for at least one year

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Mothers will participate. Child gender is a control variable.
Enrollment: 160 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Post-traumatic Stress Diagnostic Scale for the DSM-5 (PDS-5) | Change from baseline (pre-treatment) to mid-treatment at session 9 and 16 to upon completion of treatment (an average of 43 weeks) to six-month follow-up after treatment completion
  Post-traumatic Stress Diagnostic Scale for the DSM-5 (PDS-5) is a 24-item self-report measure of PTSD symptoms over the last month. Items are rated on a 5-point scale of frequency and severity ranging from 0 ("not at all") to 4 ("6 or more times a week/severe"). Higher scores indicate more severe PTSD symptoms. PDS-5 will be used to monitor change in PTSD symptoms over treatment implementation. PDS-5 is also used during the baseline to evaluate for inclusion/exclusion criteria.
Center for Epidemiological Studies-Depression (CES-D) | Change from baseline (pre-treatment) to mid-treatment at session 9 and 16 to upon completion of treatment (an average of 43 weeks) to six-month follow-up after treatment completion
  Center for Epidemiological Studies-Depression (CES-D) is a 20-item self-report measure of symptoms associated with depression, such as restless sleep, poor appetite, and feeling lonely. Items are rated on a 3-point scale ranging from 0 ("rarely or none of the time") to 3 ("most or almost all of the time"). Scores range from 0 to 60, with high scores indicating greater depressive symptoms. CES-D will be used to assess change in depression symptoms over treatment implementation.
Dyadic Parent-Child Interaction Coding System-IV (DPICS) | Change from baseline (pre-treatment) to mid-treatment at session 16 to upon completion of treatment (an average of 43 weeks) to six-month follow-up after treatment completion
  Dyadic Parent-Child Interaction Coding System-IV (DPICS) examines the quality of parent-child social interaction in three 5-minute situations: child-directed play, parent-directed play, and clean-up. Positive skills include praise, reflect, and describe, and negative skills include questions, commands, and criticisms. Observations are coded by trained DPICS scorers to produce total scores. DPICS scores allow us to track the changes in positive and negative parenting scores over treatment implementation.
New foster care removals | Every six-months for 10 years
  Data is collected through the New York State Child Welfare Registry (NYSCWR) semi-annually on the number of out-of-home placements for 10 years for completers and non-completers who have consented into the study. Number of new foster care removals are located by unique NYSCWR identifiers collected at time of consent. Out-of-home placement data, in addition to new substantiated welfare reports, will be used to assess recidivism.
New child abuse/neglect welfare reports | Every six-months for 10 years
  Data is collected through the New York State Child Welfare Registry (NYSCWR) semi-annually on the number of substantiated abuse/neglect reports for 10 years for completers and non-completers who have consented into the study. Number of new substantiated reports are located by unique NYSCWR identifiers collected at time of consent. New substantiated welfare reports, as well as out-of-home placement data, will be used to assess recidivism.
Family Preservation Services Usual Care (FPSUC) reports | Throughout study completion, an average 43 weeks
  Family Preservation Services Usual Care (FPSUC) is extracted from electronic records that agencies use to document services. FPSUC details the number of services accessed in preventative agencies for clients. Data will be used to statistically control for FPSUC.

SECONDARY OUTCOMES:
Structured Clinical Interview for DSM-5 (SCID-5) | Change from baseline (pre-treatment) to mid-treatment at session 16 to upon completion of treatment (an average of 43 weeks) to six-month follow-up after treatment completion
  Structured Clinical Interview for DSM-5 (SCID-5) is the gold standard for determining DSM-5 Axis I current diagnoses and psychiatric history. The SCID-5 alcohol and substance use and psychosis modules will be used. SCID-5 will be used to track changes in substance use/abuse and symptoms of psychosis, as well as to evaluate inclusion/exclusion criteria.
Difficulties in Emotion Regulation Scale (DERS) | Change from baseline (pre-treatment) to mid-treatment at session 9 and 16 to upon completion of treatment (an average of 43 weeks) to six-month follow-up after treatment completion
  Difficulties in Emotion Regulation Scale (DERS) is a 36-item self-report measure used to assesses emotion regulation. Items are rated on a scale of 1 ("almost never [0-10%]") to 5 ("almost always [91-100%]"). Higher scores indicate more difficulty in emotion regulation. DERS has adequate construct and predictive validity and good test-retest reliability. DERS will be used to evaluate level of emotion regulation skills during treatment implementation.
Adult Adolescent Parenting Inventory-2.1 (AAPI-2.1) | Change from baseline (pre-treatment) to end of treatment (average 43 weeks) to six-month follow-up
  Adult Adolescent Parenting Inventory-2.1 (AAPI-2.1) is a self-reporting inventory that measures parental behaviors and is commonly used to assess the risk of child abuse and neglect. Items are rated on a scale of 1 ("strongly agree") to 5 ("strongly disagree"). AAPI-2.1 has five sub-constructs: expectations of children, parental empathy towards children's needs, use of corporal punishment, parent-child family roles, and children's power and independence. Higher scores indicate lower risk of parental abuse/neglect. AAPI will be used to monitor the change in parental behaviors over treatment implementation.
Treatment Services Review (TSR) | Baseline (pre-treatment)
  Treatment Services Review (TSR) is an interview used to gather information about specific mental health services received outside of the study treatment and treatment received one year prior to the time of the baseline (pre) assessment. It describes treatment type (individual therapy vs. group), provider type (psychologist, psychiatrist, social worker), length (in years) and frequency of treatment (rate of appointments), rate of hospitalizations, and medications prescribed.
Treatment Services Review (TSR) | End of treatment (an average 43 weeks)
  Treatment Services Review (TSR) is an interview used to gather information about specific mental health services received outside of the study treatment and treatment received during treatment implementation. It describes treatment type (individual therapy vs. group), provider type (psychologist, psychiatrist, social worker), length (in years) and frequency of treatment (rate of appointments), rate of hospitalizations, and medications prescribed.
Treatment Services Review (TSR) | Follow-up after treatment completion (six-months after end of treatment)
  Treatment Services Review (TSR) is an interview used to gather information about specific mental health services received outside of the study treatment and treatment received between the end of treatment and the six-month follow-up assessment. It describes treatment type (individual therapy vs. group), provider type (psychologist, psychiatrist, social worker), length (in years) and frequency of treatment (rate of appointments), rate of hospitalizations, and medications prescribed.
Therapy Acceptability and Expectations (TAE) | Change from baseline (pre-treatment) to mid-treatment at session 9 and 16 to upon completion of treatment (an average of 43 weeks) to six-month follow-up after treatment completion
  Therapy Acceptability and Expectations (TAE) is a 5-item scale that evaluates credibility and engagement of study treatment. Items range from 0 ("not at all") to 8 ("extremely"). Higher scores indicate greater acceptability of treatment. TAE is administered throughout treatment in order to assess the clinician-client therapeutic relationship and client engagement with treatment. Necessary changes that arise from the TAE are addressed in future treatment sessions.
Strengths and Difficulties Questionnaire (SDQ) | Change from baseline (pre-treatment) to mid-treatment at session 9 and 16 to upon completion of treatment (an average of 43 weeks) to six-month follow-up after treatment completion
  Strengths and Difficulties Questionnaire (SDQ) is a 25-item parent-report behavioral screening questionnaire that comprises five sub-scales: emotional symptoms, conduct problems, hyperactivity/inattention, peer relationship problems, and prosocial behavior. Items have the following responses: "not true," "somewhat true," and "certainly true." Higher scores indicate a higher likelihood of emotional and/or behavioral difficulties. SDQ will be used throughout treatment to assess change in behavior of the child participating in the parent-child dyadic play observations.
Working Alliance Inventory Short Form (WAI-S) | Change from mid-treatment at session 9 and 16 to upon completion of treatment (an average of 15 weeks).
  The WAI-S is a 12-item measure assessing three key aspects of the therapeutic alliance: agreement on the tasks of therapy, agreement on the goals of therapy, and development of an affective bond. Item responses range from 1 ("Never") to 7 ("Always"). Higher scores indicate a higher quality of the therapeutic alliance. The WAI-S is administered throughout treatment beginning at mid-treatment in order to assess the working relationship between a client and their treating clinician, from both the participant and clinician perspectives.

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Lindsey, Principal Investigator — New York University
Locations (1):
- McSilver Institute for Poverty Policy and Research, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Informed Consent Form (2025-09-18): https://cdn.clinicaltrials.gov/large-docs/18/NCT04752618/ICF_000.pdf